CLINICAL TRIAL: NCT01998672
Title: A Double-blind, Randomised, Placebo-controlled, Dose-escalation Study of the Safety, Tolerability and Pharmacokinetics of Increasing Multiple Oral Doses of Px-102 to Healthy Subjects
Brief Title: Multiple Ascending Oral Dose Phase I Study With Px-102
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Phenex Pharmaceuticals AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PHS-Px-102-I-02
Record Dates: First submitted 2013-11-19; First posted 2013-12-02 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Healthy
MeSH Terms: interventions — PX-102

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Px-102 (Active Comparator): Px-102 drinking solution, 0.5 mg/kg, 1.0 mg/kg and 1.5 mg/kg
  Interventions: Drug: Px-102
- Placebo (Placebo Comparator): Oral drinking solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Px-102 — Px-102 drinking solution, 0.5 mg/kg, 1.0 mg/kg and 1.5 mg/kg
  Arms: Px-102
Drug: Placebo — Drinking solution
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and tolerability of the FXR agonist Px-102 in healthy subjects after 7 days multiple oral dosing.

DETAILED DESCRIPTION:
The study is a single-centre, double-blind, randomized, placebo-controlled, parallel group phase I study with healthy male subjects receiving ascending multiple oral oral doses of Px-102 to assess the safety and tolerability, pharmacokinetics and pharmacodynamics.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subject of Caucasian origin 18 to 45 years of age (inclusive).
* Good state of health (mentally and physically) as determined by medical history, physical examination, vital signs, ECG recording and clinical lab results.
* BMI in between 20-29 kg/m² (inclusive); with absolute weight in between 70 to 120 kg.
* Total cholesterol and liver enzyme levels [alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma-glutamyltransferase (GGT), alkaline phosphatase (AP)] strictly within the normal ranges at screening and on Day -1. Serum triglyceride not exceeding the upper limit of normal range.
* HbA1c ≤ 6.5%
* Subject has been informed both verbally and in writing and has given written consent to participation in the study prior to start and any study-related procedure.
* Negative results for HIV- and Hepatitis-B and -C serology at screening.
* Subject (including female partners of childbearing potential) has to use a highly effective method of birth control (failure rate less than 1% per year when used consistently and correctly), e.g. implants, injectables, combined oral contra-ceptives in combination with a barrier method, some intrauterine contraceptive devices or sexual abstinence.

Exclusion Criteria:

* Female gender
* Use of prescription or non-prescription drugs within 7 days (30 if the drug is a possible enzyme inducer) prior to administration of study medication. Use of drugs known to induce steatosis (e.g. valproate, amiodarone or prednisone) or to affect body weight and carbohydrate metabolism
* Any acute or chronic illness or clinically relevant finding at screening and at base-line examination which may jeopardize the subject's participation in the study
* History or presence of biliary obstruction or biliary disease, hepatic encephalopathy, advanced ascites, portal hypertension, esophageal/gastric variceal bleeding, hepatocellular carcinoma, previous liver transplantation or any other chronic liver disease
* Renal dysfunction, e.g. glomerular filtration rate ≤ 80 ml/min/1.73 m2 (as determined by the formula of Cockroft-Gault)
* Type I or II Diabetes
* Any clinically relevant abnormality on screening medical assessment, laboratory examination, 12-lead ECG
* Any clinically relevant finding in the baseline telemetry within the pre-dose evaluated observation period of at least 20 hours
* Marked baseline prolongation of QT/QTc interval (QTc interval > 440 ms) in the 12-lead ECG using the Fridericia method for QTc analysis
* Heart rate < 50 bpm.
* History of pathological cardiovascular symptoms or a severe cardiovascular event
* History of severe chronic autoimmune diseases such as severe allergy, atopic eczema, chronic dermatitis, severe psoriasis, multiple sclerosis, severe asthma, lupus or related disorders
* Allergies (except for mild forms of hay fever) or history of hypersensitivity reactions
* Smoking (regular or irregular) > 5 cigarettes (or equivalent) per day
* Excessive alcohol drinking (more than approximately 20 g alcohol per day), unable to refrain from alcohol drinking from 48 hours prior to dosing until the last pharmacokinetic blood sample has been withdrawn
* Positive test for drugs or alcohol at screening or prior to the dosing session
* History of alcoholism or drug/chemical/substance abuse within past 2 years
* Investigator deems the subject unable or unwilling to comply fully with the study protocol
* Has received clinical study medication within the last 30 days prior to this study
* Donation or loss of 400 ml or more of blood within eight (8) weeks prior to dosing
* Allergic to any of the active or inactive ingredients in the study medication
* Any other reason which the Investigator considers unsuitable for the subject to participate
* Any condition or previous disease leading to pruritus or itching of the skin.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2012-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of Px-102 | 7 days
  Adverse event monitoring, laboratory values, cardiovascular monitoring. Comparison active vs. placebo

SECONDARY OUTCOMES:
Pharmacokinetics of Px-102 and metabolites | Day 1: 0 min, 15 min, 30 min, 60 min, 1.5 h, 2 h, 3 h, 4 h, 5 h, 6 h, 7 h, 8 h, 12 h, 22 h, 24 h; Day 5 and 6: pre-dose; Day 7: 0 min, 15 min, 30 min, 60 min, 1.5 h, 2 h, 3 h, 4 h, 5 h, 6 h, 7 h, 8 h, 12 h, 22 h, 24 h, 30 h.
  Plasma, urine and fecal concentrations (ng/mL) of Px-102 and metabolites measured by LC-MS/MS. AUC, Cmax and other pk parameters. Comparison of the pk data on day 7 vs. day 1
Pharmacodynamics | Pre-dose, 1, 2, 4, 8 and 10 hours after administration on Days 1 and 7; Pre-dose, 2 hours and 8 hours after administration on Days 2 to 6; at 22 hours after the last administration
  Markers for FXR activation (e.G. FGF19 (pg/mL) measurement by ELISA). Comparison active vs. placebo

CONTACTS AND LOCATIONS:
Overall Officials: Claus Kremoser, Dr., Study Chair — Phenex Pharmaceuticals AG
Locations (1):
- FOCUS Clinical Drug Development GmbH, Neuss, Germany